CLINICAL TRIAL: NCT02392832
Title: Impact and Cost-Effectiveness of Long-Lasting Microbial Larvicides in Reducing Malaria Transmission and Clinical Malaria Incidence: a Cluster-Randomized Controlled Trial in Western Kenya
Brief Title: Evaluation of Long-Lasting Microbial Larvicides in Reducing Malaria Transmission and Clinical Malaria Incidence
Acronym: LLML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: R01A1050243 [HS# 2008-6148]
Record Dates: First submitted 2015-02-03; First posted 2015-03-19 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Malaria
Keywords: long-lasting microbial larvicide; intervention; cluster randomised controlled trial; Anopheles mosquito
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): Fourstar® granule formulation, 90day and 180 day briquettes Bti/Bs in larval habitats of malaria vectors.
  Interventions: Biological: Fourstar® granule, 90 day and 180 day briquettes Bti/Bs
- Control arm (No Intervention): No larvicide application.

INTERVENTIONS:
Biological: Fourstar® granule, 90 day and 180 day briquettes Bti/Bs — In 2015: Two sites each in Kakamega and Vihiga counties in western Kenya will be randomly selected and treated with larvicides (intervention) and the other two sites will serve as control (no-intervention). Temporary habitats will be treated with FourStar® controlled release granule formulation, semi-permanent habitats will be treated with 90 day briquettes, and permanent habitats with 180 day briquettes. No retreatment.
  Starts from 2016, a total of 34 clusters in the two study sites will be assigned to treatment or control by a block randomization method. The Bti treatment will be the same as in 2015. The retreatment interval will be 4-5 months. After the third treatment, no treatment will be performed for the next 8 months. After this, a cross over will be performed. Previous control sites will receive 3 rounds of the same LLML treatment at appropriate time intervals and previous treatment sites will not receive any LLMLs.
  Arms: Intervention arm

SUMMARY:
In the past decade, massive scale-up of insecticide-treated nets (ITN) and indoor residual spraying (IRS), together with the introduction of artemisinin-combination treatments, have led to substantial reductions in malaria prevalence and incidence in African highlands. However, rising insecticide resistance and increased outdoor transmission have greatly hampered the effectiveness of ITN and IRS because the current indoor-based interventions do not target the outdoor-biting mosquitoes. Therefore, new supplemental interventions that can tackle outdoor transmission and pyrethroid insecticide resistance are urgently needed. The central objective of this study is to determine the efficacy and cost-effectiveness of EPA-approved long-lasting microbial larvicides in reducing malaria transmission and clinical malaria incidence in western Kenya highlands.

DETAILED DESCRIPTION:
In the past decade, massive scale-up of insecticide-treated nets (ITNs) and indoor residual spraying (IRS), together with the use of artemisinin combination treatments, have led to major changes in malaria epidemiology and vector biology. Along with the significant reduction in overall malaria prevalence and incidence, extensive use of insecticides has created large selection pressures for resistance in the malaria vector populations and for potential outdoor transmission, which appears to be limiting the success of ITNs and IRS. Because IRS and ITN have little impact on outdoor resting and early biting vectors, outdoor transmission represents one of the most important challenges in malaria control. Therefore, new interventions that can augment the current public health measures to reduce outdoor transmission are urgently needed. Larval control has historically been very successful and is widely used for mosquito control in many parts of the world, except in Africa. Factors limiting the use of larvicides include high costs associated with frequent habitat re-treatment. Now a new US EPA-approved long-lasting formulation, potentially effective for 6 months is available. The central objective of this study is to determine the effect of long-lasting microbial larviciding on the incidence of clinical malaria and reduction of transmission intensity. Our hypothesis is that addition of long-lasting microbial larviciding to ongoing ITN and IRS programs will lead to significant reductions in both indoor and outdoor malaria transmission and malaria incidence.

ELIGIBILITY:
Inclusion Criteria:

* All clinical malaria cases from participated local hospitals and clinics.

Exclusion Criteria:

* Infants younger than 6 months.

Min Age: 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240000 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Changes in clinical malaria incidence rate | baseline and 4 months following the interventions
  Human population for each site stratified into three age groups, under 5 years, 6-15 years and >15 years, will be ascertained from our existing demographic database. Age group level aggregate morbidity data with number of clinical malaria cases without any identifiers will be obtained from local hospitals and clinics where the study residents seek treatment. This data is reported to the Ministry of Health of Kenya and hence, is publicly available.

SECONDARY OUTCOMES:
Changes in vector abundance | baseline and 4 months following the interventions
  Malaria vector abundance is measured by the total density of An. gambiae, An. arabiensis, An. funestus and other Anopheles species capable of transmitting malaria, collected indoors and outdoors by the CO2-baited CDC light trap, 64 trap nights in each of indoor and outdoor environments per site per month. Malaria transmission intensity is measured by the sum of indoor and outdoor entomological inoculation rate (EIR).
EIR | baseline and 4 months following the interventions
  Malaria transmission intensity is measured by the sum of indoor and outdoor entomological inoculation rate (EIR).

CONTACTS AND LOCATIONS:
Overall Officials: Guiyun Yan, Ph.D., Principal Investigator — University of California at Irvine
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
We use aggregated publically available clinical records from hospitals, these records can be obtained freely from hospitals or Ministry of Health. We can provide these aggregated data upon request once they are published.
Time Frame: Will be available by June 30, 2020
Access Criteria: Available to public

REFERENCES:
- [Derived] Zhou G, Wiseman V, Atieli HE, Lee MC, Githeko AK, Yan G. The impact of long-lasting microbial larvicides in reducing malaria transmission and clinical malaria incidence: study protocol for a cluster randomized controlled trial. Trials. 2016 Aug 25;17(1):423. doi: 10.1186/s13063-016-1545-4. PMID 27558161